CLINICAL TRIAL: NCT02495584
Title: D-Light Intervention: A Randomised Controlled Human Intervention Study to Assess the Impact of Vitamin D From Milk and Supplements on Functional Health Outcomes and Future Vitamin D Synthesis From UV Exposure
Brief Title: D-Light Intervention
Acronym: D-Light
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Dairy Council for Northern Ireland (Other); Agri-Food and Biosciences Institute (Other); Center for Nutrition and Health, RIVM (The Netherlands) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 13/NI/0091
Record Dates: First submitted 2015-05-11; First posted 2015-07-13 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: 25-hydroxyvitamin D Concentration (Vitamin D Status)
Keywords: Vitamin D; Fortified milk; Supplementation; UV exposure; Winter; Healthy adults; Body Composition; Muscle function; Blood pressure
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment 1 (Experimental): 500ml fortified milk (10µg vitamin D3) +1 supplement capsule (10µg vitamin D3) daily for 24 weeks
  Interventions: Dietary Supplement: Fortified milk (10µg vitamin D3); Dietary Supplement: 10µg vitamin D3 supplement
- Treatment 2 (Experimental): 500ml fortified milk (10µg vitamin D3) +1 supplement capsule (placebo) daily for 24 weeks
  Interventions: Dietary Supplement: Fortified milk (10µg vitamin D3); Dietary Supplement: Placebo supplement
- Treatment 3 (Experimental): 500ml unfortified milk (placebo) +1 supplement capsule (10µg vitamin D3) daily for 24 weeks
  Interventions: Dietary Supplement: Unfortified milk (placebo); Dietary Supplement: 10µg vitamin D3 supplement
- Treatment 4 (Placebo Comparator): 500ml unfortified milk (placebo) +1 supplement capsule (placebo) daily for 24 weeks
  Interventions: Dietary Supplement: Unfortified milk (placebo); Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Fortified milk (10µg vitamin D3)
  Arms: Treatment 1; Treatment 2
Dietary Supplement: Unfortified milk (placebo)
  Arms: Treatment 3; Treatment 4
Dietary Supplement: 10µg vitamin D3 supplement
  Arms: Treatment 1; Treatment 3
Dietary Supplement: Placebo supplement
  Arms: Treatment 2; Treatment 4

SUMMARY:
Vitamin D insufficiency has become a global concern, with low vitamin D status associated with bone disorders, cardiovascular disease and certain cancers. The United Kingdom (UK) and Ireland are at particular risk of vitamin D deficiency owing to the northerly latitude, increased use of sunscreen, decreased sun exposure and a high level of cloud cover. A recent survey in the UK showed that more than 50% of UK adults have insufficient vitamin D status, with lower levels noted in the winter months. Variations in vitamin D status have been known to vary between summer and winter, owing to our northern latitude (52-55°N) the Ultraviolet (UV)-B intensity in Northern Ireland is inadequate to promote the dermal synthesis of vitamin D during the winter months, causing us to rely on dietary sources. The aim of this intervention is to investigate the main effects of vitamin D3-fortified milk and supplemental vitamin D3 on vitamin D status and functional health outcomes during the winter, and how this intervention will affect subsequent dermal synthesis of vitamin D from UV exposure. Participants will be recruited from the local community. Blood samples will be collected from each participant at two timepoints (September/October and March/April). Pre- and post-intervention blood pressure, grip strength, height, weight, waist and hip circumferences will be measured, in addition participants will undergo a dual energy x-ray absorptiometry (DXA) scan to assess body composition and bone mineral density. Information on general health, lifestyle, physical activity, dietary intake and typical behaviours in the sun will be collected. Following the dietary intervention, a subset of participants will be invited to participate in a follow-up study, examining UV exposure during the summer months, when they will wear a personal wrist dosimeter for 1 month, complete a sun dairy and provide 2 additional blood samples.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 years old
* Apparently healthy
* Living on the island of Ireland

Exclusion Criteria:

* Below 20 years and aged 40 years or above
* Not living on the island of Ireland
* Pregnant or lactating women and those planning to become pregnant
* Individuals who have been taking a vitamin D or calcium containing supplement in the previous three months
* Those with food intolerances or allergies that would affect their ability to consume study milk
* Individuals following a diet which excludes milk (e.g. vegans)
* Those with a diagnosed chronic medical condition or on prescribed medication known to effect vitamin D metabolism
* Those who are planning a sun holiday during the winter months (Oct-Mar)
* Adults with learning, or any other difficulties that would prevent them from completing the study protocol

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in vitamin D status (25-hydroxyvitamin D serum concentration) | Baseline + post-intervention (24weeks)
  Blood analysis

SECONDARY OUTCOMES:
Change in body composition | Baseline + post-intervention (24weeks)
  Assessed by dual energy X-ray absorptiometry (DXA)
Change in muscle strength | Baseline + post-intervention (24weeks)
  Assessed by grip strength
Change in inflammation status | Baseline + post-intervention (24weeks)
  Blood analysis
Change in lipid profile | Baseline + post-intervention (24weeks)
  Blood analysis
Change in glucose levels | Baseline + post-intervention (24weeks)
  Blood analysis
Change in insulin concentrations | Baseline + post-intervention (24weeks)
  Blood analysis

OTHER OUTCOMES:
UV exposure (follow-up) | 8 weeks post-intervention (32-40 weeks)
  Assessed by UV wrist monitors

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Coleraine, United Kingdom